CLINICAL TRIAL: NCT01138085
Title: A Phase I Dose Escalation Open-Label Safety, Pharmacokinetic and Pharmacodynamic Study to Determine the Recommended Phase II Dose of GSK1120212 Dosed in Combination With GSK2141795
Brief Title: Safety, Pharmacokinetics (PK) of AKT and MEK Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113886
Record Dates: First submitted 2010-04-22; First posted 2010-06-07 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: Triple negative breast cancer; BRAF wild-type melanoma; Solid tumors; Endometrial Cancer; Oncology; GSK2141795; AKT Inhibitor; GSK1120212
MeSH Terms: conditions — Neoplasms; Triple Negative Breast Neoplasms; Endometrial Neoplasms | interventions — trametinib; GSK2141795

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Escalation (Experimental): Dose escalation will proceed until unacceptable toxicity is observed. Dose escalation decisions will take into account all available data, including PK data and the safety profile of prior cohorts and will occur following review of these data by the investigator(s), GSK medical monitor, pharmacokineticist, and statistician.
  Interventions: Drug: GSK1120212; Drug: GSK2141795
- Expansion Cohorts (Experimental): Enrollment into expansion cohort(s) in Part 2A may begin once a recommended dosing regimen(s) is identified in Part 1A utilizing a once daily continuous dosing schedule for both GSK1120212 and GSK2141795. Enrolment to cohorts utilizing this daily dosing schedule may proceed in parallel with enrolment in Part 1B. Expansion cohort(s) will preferentially enroll subjects with treatment-refractory, measurable and biopsiable triple negative breast cancer or BRAF- wild type melanoma. Subjects selected for enrollment into Part 2A or Part 2B will be tested for PTEN deficiency and must agree to provide paired tumor biopsies (at baseline and once while on- treatment). An additional tumor biopsy at the time of disease progression should also be collected if feasible.
  In Part 2A and Part 2B, up to 35 additional subjects per tumor type and schedule (i.e., a total of up to 70 subjects per schedule tested) may be enrolled in a two-stage design to better characterize safety, PK and PD.
  Interventions: Drug: GSK1120212; Drug: GSK2141795

INTERVENTIONS:
Drug: GSK1120212 — MEK inhibitor
Drug: GSK2141795 — AKT Inhibitor

SUMMARY:
This study is a Phase 1 dose-escalation open-label study to determine the recommended Phase II dose (RP2D) and regimen for the combination of the orally administered MEK inhibitor GSK1120212 and the orally administered AKT kinase inhibitor GSK2141795. The study consists of two parts. Part 1A will identify the maximum tolerated dose (MTD) using a Zone-Based, modified 3 plus 3 dose escalation procedure. The starting dose (Zone 1, Cohort 1) will be 0.5mg GSK1120212 combined with 25mg GSK2141795. Dose escalation will continue based on predefined parameters until a MTD is established. The initial regimen for dose escalation in Part 1A will be continuous oral daily dosing. Once the continuous daily dosing MTD or RP2D has been established in Part 1A, Part 1B will explore alternate dosing schedule(s) in which the dosing schedule may be adjusted for either GSK1120212 or GSK2141795. Dose escalation will proceed using a 3 plus 3 dose escalation procedure until an MTD or RP2D of that alternate schedule is defined. Part 2 will explore further in specific tumor types the safety, tolerability, clinical activity, pharmacokinetic (PK) and pharmacodynamic (PD) properties of the combination of GSK1120212 and GSK2141795 at the recommended dose(s) and regimen(s) identified in Part 1.

ELIGIBILITY:
Inclusion Criteria:

Part 1 - Dose Escalation

Subjects eligible for enrollment in the study must meet all of the following criteria:

Male or female 18 years or older, at the time of signing the informed consent.

Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Histologically or cytologically-confirmed diagnosis of solid tumor malignancy that is not responsive to standard therapies or for which there is no approved or curative therapy or for subjects who refuse standard therapy (Part 1A). Part 1B subjects must have a confirmed diagnosis of one of the following (documented lab results confirming mutational status must be available at Screening):

colorectal cancer (CRC): KRAS mutation non-small cell lung (NSCLC): KRAS mutation Pancreatic: no mutational status specified Endometrial: no mutational status specified Ovarian: no mutational status specified Squamous cell carcinoma of the head and neck: no mutational status specified BRAF wild type melanoma (preferentially enrolled to Part 2) BRAF inhibitor failure melanoma. This includes BRAF-mutant melanoma that is either initially refractory to BRAF-inhibitor therapy OR that Initially responds to BRAF-inhibitor therapy but eventually develops documented radiographic progression to a BRAF inhibitor while on therapy Triple negative breast cancer (TNBC) (preferentially enrolled to Part 2) NOTE: Subjects who do not meet one of the categories described above but who have molecular evidence suggesting benefit from the study drugs may be considered for enrollment after discussion with the GlaxoSmithKline (GSK) Medical Monitor.

Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.

Able to swallow and retain oral medication.

Must agree to collection of blood samples for the evaluation of circulating free DNA (cfDNA) (Part 1B or Part 2).

A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] greater than 40 MlU/ml and estradiol less than 40 pg/ml [less than 140 pmol/L] is confirmatory). Females on hormone replacement therapy [HRT] and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

Child-bearing potential and agrees to use one of the contraception methods listed in Section 7.3.2 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Additionally, women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to the first dose of study medication. Female subjects must agree to use contraception until four weeks after the last dose of study medication.

Note: Oral contraceptives are not reliable due to potential drug-drug interaction and should only be used in combination with the alternative methods outlined in Section 8.1.1.

Male subjects must agree to use one of the contraception methods listed in Section 8.1.2. This criterion must be followed from the time of the first dose of study medication until four months after the last dose of study medication.

Adequate organ system function as defined in protocol. Absolute neutrophil count (ANC) greater than or equal to 1.5 X 10 to the ninth/L Hemoglobin greater than or equal to 9.5 g/dL Platelets greater than or equal to 75 X 10 to the ninth/L Prothrombin time (PT) / International Normalized Ratio (INR) and Partial Thromboplastin Time (PTT) less than or equal to 1.1 X ULN Total bilirubin less than or equal to 1.5 x ULN (isolated bilirubin greater than 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35 percent) AST and ALT less than or equal to 1.5 X ULN Albumin greater than 2.5 g/dL Creatinine less than or equal to ULN OR Calculated creatinine clearance greater than or equal to 30 mL/min OR 24-hour urine creatinine clearance greater than or equal to 30 mL/min

Fasting Serum Glucose les than 126mg/dL Cardiac Ejection fraction greater than or equal to lower limit of normal (LLN) by ECHO

Inclusion Criteria for Part 2 - Expansion Cohort:

Histologically- or cytologically-confirmed diagnosis of one of the following:

Triple negative (estrogen receptor(ER)-/ progesterone receptor(PR)-/ human epidermal growth factor receptor 2 (HER2)) breast cancer in the locally advanced or metastatic setting BRAF-wild type melanoma. Based on emerging data, subjects with these tumor histologies may be required to meet specific genetic selection criteria if those criteria are felt to improve the likelihood that a given subject will respond to study drug(s). If this is to occur, the site and the Investigational Review Board (IRB) will be notified but this change will not constitute a protocol amendment.

Known Phosphatase and tensin homolog (PTEN) status of tumor. At least 6 of the subjects enrolled in Stage 1 with each tumor type will have PTEN deficiency while at least 6 others will be PTEN wild type.

If the subject's tumor PTEN status was previously determined by an acceptable, analytically validated assay (i.e., Immunohistochemistry (IHC), fluorescence in situ hybridization (FISH), sequencing, copy number analysis) then PTEN by IHC at Screening will not need to be repeated for the purpose of enrollment in this study. However, archival tumor tissue or tissue from a fresh biopsy specimen should be submitted for confirmation of PTEN status by a central laboratory using IHC.

If PTEN status was not previously determined, archival tissue from a previous tumor biopsy specimen must be available for PTEN IHC analysis; if archival tissue is not available or found to not contain tumor tissue, a fresh biopsy is required to obtain tumor tissue for testing.

Subjects in Part 2 that have been previously diagnosed with Type 2 diabetes must also meet the additional following criteria:

Diagnosis of diabetes greater than or equal to 6 months prior to enrolment HbA1C less than or equal to 8 percent at Screening visit

Exclusion Criteria

Subjects meeting any of the following criteria must not be enrolled in the study:

Chemotherapy, radiotherapy, immunotherapy, or other anti-cancer therapy including investigational drugs within 28 days or 5 half lives, whichever is shorter prior to the first dose of any one of the investigational drugs described in this study. Prior exposure to either a MEK inhibitor or an AKT inhibitor is not permitted.

Current use of a prohibited medication or requires any of these medications during treatment with the study treatments.

Unresolved toxicity greater than National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 (NCI-CTCAE v4) Grade 1 from previous anti-cancer therapy unless agreed to by a GSK Medical Monitor and the Investigator, and where a GSK Medical Monitor and the investigator consider that the ongoing toxicity will not introduce additional risk factors and will not interfere with the study procedures.

Presence of active gastrointestinal (GI) disease or other condition that could affect gastrointestinal absorption (e.g. malabsorption syndrome) or predispose a subject to GI ulceration. Subjects with prior Whipple procedure are eligible.

Evidence of mucosal or internal bleeding.

Any major surgery within the last four weeks.

Previously diagnosed with Type 1 diabetes mellitus.

Previously diagnosed with Type 2 diabetes (Part 1A or Part 1B ONLY). Subjects with a history of steroid-induced hyperglycemia may be enrolled.

Any malignancy related to human immunodeficiency virus (HIV), history of HIV, history of known hepatitis B virus (HBV) surface antigen positivity (subjects with documented laboratory evidence of HBV clearance may be enrolled) or positive hepatitis C virus (HCV) antibody.

Known active infection requiring parenteral or oral anti-infective treatment.

Subjects with leptomeningeal disease.

Subjects with brain metastases are excluded if their brain metastases are:

Symptomatic Treated (e.g., surgery, radiation therapy) but not clinically and radiographically stable one month after therapy (as assessed by at least two distinct contrast enhanced magnetic resonance imaging (MRI) or computerized axial tomography (CT) scans over at least a one month period), OR Asymptomatic and untreated but greater than 1 cm in the longest dimension Subjects with small (less than or equal to 1 cm in the longest dimension), asymptomatic brain metastases that do not need immediate therapy can be enrolled. Subjects must also be off of enzyme-inducing anticonvulsants for more than 4 weeks.

Part 1B: Subjects with brain metastases who have been off corticosteroids for at least 2 months can be enrolled.

Part 2 (A or B): Subjects with brain metastases on a stable (i.e., unchanged) dose of corticosteroids for more than one month, or those who have been off corticosteroids for at least 2 weeks can be enrolled.

QTcF interval greater than or equal to 480 milliseconds (msecs) (greater than or equal to 500 msec for subject with bundle branch block).

History or evidence of current clinically significant uncontrolled arrhythmias. Subjects with controlled atrial fibrillation for greater than 1 month prior to study Day 1 are eligible.

History of acute coronary syndromes (including unstable angina), myocardial infarction, coronary angioplasty, or stenting or bypass grafting within six months of Screening.

Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.

Other clinically significant electrocardiography (ECG) abnormalities including 2nd degree (Type II) or 3rd degree atrioventricular (AV) block.

Subject with intra-cardiac defibrillators or pacemaker.

Presence of cardiac metastases.

Any serious or unstable pre-existing medical, psychiatric, or other condition (including lab abnormalities) that could interfere with subject's safety or providing informed consent.

Known immediate or delayed hypersensitivity to any of the components of the study treatment(s).

Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease, including unstable hypertension).

Pregnant or lactating females.

History or current evidence / risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR):

History of RVO or CSR, or the presence of predisposing factors to RVO or CSR at the time of screening (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes).

Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or CSR such as:

Evidence of new optic disc cupping Evidence of new visual field defects Intraocular pressure greater than 21 mm Hg as measured by tonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-05-04 (Actual); Primary Completion 2014-11-19 (Actual); Study Completion 2014-11-19 (Actual)

PRIMARY OUTCOMES:
Part 1A: To determine the safety, tolerability and recommended Phase II dose of GSK1120212 and GSK2141795 administered in combination orally, once daily continuously | Duration of study.
Part 1B:To determine the safety, tolerability and recommended Phase II dose of GSK1120212 and GSK2141795 administered in combination with an alternate schedule (i.e., at least one agent is dosed intermittently) | Duration of study
Parts 2A/2B: To evaluate the clinical activity of GSK1120212 and GSK2141795 administered in combination in subjects with solid tumors that are predicted to be sensitive to the inhibition of MEK and/or AKT, including TNBC and BRAF-wild type melanoma | Duration of study

SECONDARY OUTCOMES:
To characterize the PK of GSK1120212 and GSK2141795 for a once daily continuous dosing schedule (Part 1A) and/or an intermittent dosing schedule (Part 1B). | duration of study
Part 1A, Part 1B: To evaluate the clinical activity of GSK1120212 and GSK2141795 in subjects with solid tumors. | Duration of study
Parts 1 and 2: To characterize the durability of response with GSK1120212 and GSK2141795 dosed orally in combination | Duration of study
To evaluate the pharmacodynamic (PD) response in tumors after treatment with the combination of GSK1120212 and GSK2141795. | Duration of study
To explore relationships between study drug PK, PD and clinical activity | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (9):
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah

REFERENCES:
- See also: Results for study 113886 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113886?search=study&search_terms=113886#rs